CLINICAL TRIAL: NCT00018161
Title: Combined Pharmacologic/Behavioral Treatment for Smoking Cessation
Brief Title: Treatment to Quit Smoking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADRD-008-97F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-09

CONDITIONS: Smoking
Keywords: Nicotine; addiction; cigarette smoking
MeSH Terms: conditions — Smoking; Behavior, Addictive; Cigarette Smoking | interventions — Mecamylamine; Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: Mecamylamine
Drug: Nicotine Patch
Behavioral: Cigarette brand switching

SUMMARY:
This protocol evaluates the efficacy of combining pharmacologic treatments for smoking cessation, entailing the use of the nicotine skin patch with the nicotinic antagonist mecamylamine, with a specific behavioral therapy designed to inhibit the smoking urge.

DETAILED DESCRIPTION:
Previous studies have found that nicotine/mecamylamine treatment more than doubles the long-term abstinence rates relative to nicotine replacement alone. Recent evidence supports the hypothesis that nicotine/mecamylamine treatment prior to smoking cessation partially blocks the rewarding effects of cigarette smoking and hence promotes extinction of the smoking habit, facilitating subsequent abstinence. The behavioral approach employed is also an extinction strategy and involves having smokers switch to de-nicotinized tobacco cigarettes for two weeks prior to quitting smoking. It is hypothesized that the use of de-nicotinized cigarettes might provide more complete extinction than provided by the partial pharmacologic blockade using nicotine/mecamylamine alone. The pharmacologic treatment was expected to increase compliance with the de-nicotinized cigarette smoking regimen, because subjects' usual brands of cigarettes will be less appealing than in the absence of nicotine/mecamylamine treatment. Together the brand-switching and nicotine/mecamylamine therapies were expected to reduce cravings and other withdrawal symptoms as well as increase long-term abstinence from smoking.

ELIGIBILITY:
* Smokers,
* Ages 18-65, wanted to quit smoking.
* Must be in good health
* Exclude cardiac disease, hypotensive or hypertensive, skin allergy, glaucoma, prostatic hypertrophy, pregnant women, drug or alcohol abuse, kidney disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-01; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Westman, M.D.
Locations (1):
- Veterans Affairs Medical Center, Durham, North Carolina, United States